CLINICAL TRIAL: NCT05708573
Title: A Phase 1 Study to Evaluate the Potential Drug Interaction Between ALXN2040 and Rosuvastatin in Healthy Adult Participants
Brief Title: Potential Drug Interaction Between ALXN2040 and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN2040-HV-102
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Healthy Participants
Keywords: Drug-drug interaction; Breast cancer resistance protein; organic-anion transporting polyprotein
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Participants will receive a single dose of rosuvastatin in the morning of Day 1 in Treatment Period 1. Following a washout period of 5 days, participants will receive ALXN2040 three times daily on Days 1 through 7 in treatment period 2.
  Interventions: Drug: Rosuvastatin; Drug: ALXN2040

INTERVENTIONS:
Drug: Rosuvastatin — In Treatment Period 1, participants will receive a single oral tablet of rosuvastatin in the morning of Day 1. In treatment period 2, on the morning of Day 4, participants will receive a single 20 mg dose of rosuvastatin (co-administered with the morning dose of ALXN2040).
Drug: ALXN2040 — In Treatment Period 2, participants will receive oral tablets of ALXN2040 three times daily on Days 1 through 7.

SUMMARY:
This study will assess the potential drug-drug interaction (DDI) between ALXN2040 and rosuvastatin.

DETAILED DESCRIPTION:
This is an open-label, 2-treatment, 2-period, fixed-sequence DDI study in healthy adult participants.

This study will comprise of:

* Screening duration of 27 days.
* Two treatment periods: Approximately 14 days. Treatment Period 1: 6 days Treatment Period 2: 8 days
* Follow-up: 7 (± 2) days following the final dose of study intervention.

There will be a washout period of at least 5 days between the single dose of rosuvastatin in Treatment Period 1 and the first dose of ALXN2040 in Treatment Period 2.

Each participant will be involved in the study for approximately 48 days.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy participants with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory safety evaluation (hematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with participation in or ability to complete the study, or to potentially confound interpretation of study results, as assessed by the Investigator.
* Body mass index (BMI) within the range 18 to 32 kg/m^2 (inclusive), with a minimum body weight of 50.0 kg at Screening.

Exclusion Criteria:

* History of any medical or psychiatric condition or disease that, in the opinion of the Investigator, might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* History of meningococcal infection.
* History of drug or alcohol abuse within 2 years prior to first dose of study intervention, or positive drugs-of-abuse or alcohol screen at Screening or Day -1.
* Current tobacco users or smokers or a positive cotinine test at Screening.
* Any major surgery within 8 weeks of Screening.
* Donation of whole blood from 3 months prior to first dose, or of plasma from 30 days prior to first dose of study intervention.
* History of malignancy within 5 years prior to Screening.
* Evidence of human immunodeficiency virus (HIV) infection (HIV antibody positive) at Screening.
* Evidence of hepatitis B (positive hepatitis B surface antigen or positive core antibody with negative surface antibody) or hepatitis C viral infection (hepatitis C virus antibody positive) at Screening.
* Female participant who is pregnant, breastfeeding, or intending to conceive during the course of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration during a dosing interval (Cmax) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Area under the concentration-time curve from time zero to the time of the last observed/measured nonzero concentration (AUC0-last) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Time to reach Cmax (tmax) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
First-order rate constant of drug associated with the terminal portion of the curve (λz) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Percentage of AUC0-inf due to extrapolation from time of last quantifiable concentration to infinity (AUC%extrap) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Apparent volume of distribution during the terminal elimination phase after extravascular administration (Vd/F) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Apparent total plasma clearance after extravascular administration (CL/F) of rosuvastatin | Up to 96 hours postdose
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Cmax of ALXN2040 | Treatment Period 2: Days 3 and 4 (Predose and Postdose) [Treatment period 2 is of 8 days]
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
tmax of ALXN2040 | Treatment Period 2: Days 3 and 4 (Predose and Postdose) [Treatment period 2 is of 8 days]
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.
Area under the concentration-time curve from time zero to 8 hours postdose (AUC0-8) of ALXN2040 | Treatment Period 2: Days 3 and 4 (Predose and Postdose) [Treatment period 2 is of 8 days]
  To determine the effect of multiple doses of ALXN2040 on the single-dose PK of rosuvastatin.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Screening (Day -28 to -2) Up to Follow-up Visit (7 ± 2 days after the last dose of study intervention, or at early discontinuation from the study) [approximately 48 days]
  To assess the safety and tolerability of multiple doses of ALXN2040 when co administered with a single dose of rosuvastatin.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home